CLINICAL TRIAL: NCT05208515
Title: A Randomized, Standard-controlled Study of Establishing Independent Obstetric Operating Centre and Decision-to-delivery Interval for Emergency Cesarean Section
Brief Title: The Effect of Independent Obstetric Operating Room on Decision-to-delivery Interval for Emergency Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maternal and Child Health Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Zhengping Liu, MD, Director, Maternal and Child Health Hospital of Foshan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCHHFoshan-2199
Record Dates: First submitted 2021-12-23; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Emergency Cesarean Section
Keywords: independent obstetric operating room; emergency cesarean section; decision-to-delivery interval

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stardard group (Other): wowen who need emergency cesarean section will be send to the general operating center.
  Interventions: Other: general operating center
- new group (Experimental): women who need emergency cesarean section will be send to the obstetric operating center
  Interventions: Other: independent obsteric operating center

INTERVENTIONS:
Other: independent obsteric operating center — send emergency cesarean section needing women from labor room to independent obstetric operating center
  Arms: new group
Other: general operating center — send emergency cesarean section needing women from labor room to general operating center
  Arms: stardard group

SUMMARY:
The study is to investigate whether the establishing independent obstetric operating centre can shorten the decision-to-delivery interval and improve delivery outcomes of emergency cesarean section.

DETAILED DESCRIPTION:
The newest define of decision-to-delivery interval (DDI) is the interval between the time at which the senior obstetrician makes the decision that a caesarean section is required and the time at which the fetus (or first fetus in the case of multiples) is delivered. The recommended DDI by the American College of Obstetricians and Gynecologists and the Royal College of Obstetricians and Gynecologists is within 30 minutes. The 30 minutes rule is also used to measure the overall performance of an obstetric unit in our country. Lower rate of DDI over 30 minutes will improve the outcome of neonatal outcomes.

Affiliated Foshan Maternity & Child Healthcare Hospital is a tertiary care hospital in south of our country. Obstetric operations in this hospital are used to perform in a big general operating center, which is shared by all departments of the hospital. In December 23, 2020, a new wing of the hospital opened in response to the growing number of patients. In the new wing, an independent obstetric operating center was established to provide health care for obstetric operating. The original and new obstetric units were built according to the same standard. The medical staff shifts between original and new obstetric units every three months. Six months after the new wing of hospital opened, we set off a randomized and controlled trial (RCT). The RCT is aimed to investigate whether the independent obstetric operating center can shorten the DDI, decrease the rate of DDI over 30 minutes and improve neonatal outcomes.

Women who are over 18 years old, meet the conditions of vaginal delivery and decided to give birth vaginally by doctor and patient will be random distributed to original or new obstetric unit from July 1, 2021 to June 30,2022. Women need ECS in original obstetric unit will be send to the general operating center (named standard group), those need ECS in the new wing will be send to the obstetric operating center (named new group). DDI and other related variables of those who need ECS will be recorded. Data of a total of 60 ECS in each group will be collected and analyzed at last. Women who with missing data should be excluded.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old, meet the conditions of vaginal delivery, decided to give birth vaginally

Exclusion Criteria:

* with missing data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
decision to delivery interval | labor day
  the interval between the time at which the senior obstetrician makes the decision that a caesarean section is required and the time at which the fetus (or first fetus in the case of multiples) is delivered.
transfer time | labor day
  Time of decision to time of arrival of the patient in theatre
anesthetic time | labor day
  Arrival of the patient in theatres to anaesthetic ready time
Operation waiting time | labor day
  Time at which the anaesthetic is ready to the first skin incision
delivery time | labor day
  Skin incision-to-delivery of the first fetus

SECONDARY OUTCOMES:
number of still birth | labor day
  number of a birth in which the baby is born dead
number of neonatal death | labor day
  number of newborn died after birth
first minute Apgar score | labor day
  Apgar score is a measure of the physical condition of a newborn infant. It is obtained by adding points (2, 1, or 0) for heart rate, respiratory effort, muscle tone, response to stimulation, and skin coloration; a score of ten represents the best possible condition. The 1-minute score determines how well the baby tolerated the birthing process.
five minutes Apgar score | labor day
  Apgar score is a measure of the physical condition of a newborn infant. It is obtained by adding points (2, 1, or 0) for heart rate, respiratory effort, muscle tone, response to stimulation, and skin coloration; a score of ten represents the best possible condition. The 5-minute score tells the health care provider how well the baby is doing outside the mother's womb.
degree of neonatal asphyxia | labor day
  neonatal asphyxia is divied into no (8~10), mild(4~7) and sever(0~3) accroding to the Apgar score evaluated in one minute.
number of newborn transferred to NICU | From delivery to one week after delivery
  number of newborn transferred to neonatal intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Maternal and Child Health Hospital of Foshan, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No